CLINICAL TRIAL: NCT02428270
Title: Molecular Basket Trial In Multiple Malignancies With Common Target Pathway Aberrancies: A Phase II Trial of GSK2256098 and Trametinib in Patients With Advanced Pancreatic Cancer
Brief Title: A Study of GSK2256098 and Trametinib in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOBILITY-002
Record Dates: First submitted 2015-04-23; First posted 2015-04-28 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer; Adenocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — GSK2256098; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GSK2256098 and Trametinib (Experimental): GSK2256098, orally, at 0.375 or 0.5 mg, once daily, continuously every 28 day cycles.
  Trametinib, orally at 250 mg or 500 mg, twice daily, continuously every 28 day cycles.
  Interventions: Drug: GSK2256098; Drug: Trametinib

INTERVENTIONS:
Drug: GSK2256098 — Small molecule inhibitor of focal adhesion kinase (FAK)
Drug: Trametinib — Allosteric inhibitor of mitogen-activated extracellular signal-regulated kinase (MEK)1 and MEK2 activation and kinase activity.
  Other Names: Mekinist

SUMMARY:
This is a phase 2 study (the second phase in testing a new drug or combination to see how effect the drug or combination is) of investigational drugs GSK2256098 and Trametinib.

The purpose of the study is to evaluate the antitumor activity of GSK2256098 and Trametinib in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
Trametinib is a drug that works by binding to and blocking certain proteins called mitogen-activated protein kinase kinase (MEK) 1 and MEK2 from working. MEK1 and MEK2 are important proteins that contribute to the growth of cancer cells.

GSK2256098 is a drug that blocks a protein called focal adhesion kinase-1 (FAK) which is an important protein that contribute to the growth of cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older, able to give written consent
* Pancreatic adenocarcinoma that is not responsive to standard therapies or for which there is no approved or curative therapy or for patients who refuse standard therapy
* Have clinical, radiographic, or serologic progression after one prior line of chemotherapy for advanced disease. Patients who have received two or more prior lines of chemotherapy for advanced disease are not eligible.
* Performance Status score of 0 or 1
* Measureable disease by RECIST version 1.1
* Able to swallow and retain oral medication
* Have malignant disease that is amenable to biopsy and agree to collection of mandatory tumor biopsy samples.
* Agrees to use contraception
* Not pregnant
* Adequate organ system function

Exclusion Criteria:

* Chemotherapy, radiotherapy, immunotherapy, or other anti-cancer therapy including investigational drugs within 28 days or 5 half lives. No prior MEK inhibitor, RAF inhibitors or a FAK inhibitors
* Current use of a prohibited medication
* Unresolved toxicity greater than Grade 1 from previous anticancer therapy unless the ongoing toxicity will not introduce additional risk factors and will not interfere with the study procedures.
* Presence of active GI disease or other condition that could affect gastrointestinal absorption or predisposed to GI ulceration
* Evidence of mucosal or internal bleeding
* Anticoagulation with warfarin
* Major surgery within the last four weeks
* Malignancies related to HIV or HBV/HCV
* Known active infection requiring parenteral or oral anti-infective treatment
* Leptomeningeal disease.
* Brain metastases
* QTcF interval ≥ 480 msecs
* History or evidence of current clinically significant uncontrolled arrhythmias
* History of acute coronary syndromes, myocardial infarction, coronary angioplasty, or stenting or bypass grafting within six months of screening.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.
* Other clinically significant ECG abnormalities
* Intra-cardiac defibrillators.
* Presence of cardiac metastases.
* Serious or unstable pre-existing medical, psychiatric, or other condition that could interfere with patient's safety or providing informed consent.
* Known immediate or delayed hypersensitivity to any of the components of the study treatment(s).
* Evidence of severe or uncontrolled systemic diseases
* Pregnant or lactating
* History of retinal vein occlusion
* History of interstitial lung disease or pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04; Primary Completion 2017-06 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who experience complete response, partial response, or stable disease | 24 weeks

SECONDARY OUTCOMES:
Adverse events based on frequency and proportion of total patients, by system organ class and preferred term. | 2 years
Percentage of patients achieving either a complete or partial tumor response. | 2 years
Interval between the date of randomization and the earliest date of disease progression or death due to any cause | 2 years
Interval between the first date of CR or PR and the earliest date of disease progression or death due to any cause. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bedard, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (4):
- Canada (4):
  - Juravinski Cancer Center, Hamilton, Ontario
  - London Regional Cancer Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario